CLINICAL TRIAL: NCT06811896
Title: Adapting and Piloting a Stress Management Intervention to Reduce Cardiovascular Disease Risk Among Women Living With HIV
Brief Title: Adapting a Stress Management Intervention to Reduce Cardiovascular Disease Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jenni Wise, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300012154; 1K23HL170836-01A1 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Stress; Blood Pressure; Cardiovascular Diseases (CVD)
Keywords: stress; resiliency; meditation; blood pressure; cardiovascular risk
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Usual Care
  Interventions: Other: Usual Care
- Intervention (Other): Adapted Intervention, Previously Established
  Interventions: Behavioral: Stress Management and Resiliency Training Program

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training Program — The Stress Management and Resiliency Training Intervention is an evidence-based intervention to reduce physiologic responses to stress that may contribute to cardiovascular disease risk. The intervention is typically delivered over an 8-week period and works to decrease stress responses by improving psychological resiliency to structural and social stressors and decreasing sympathetic nervous system activation. Eliciting the relaxation response through meditation, mindfulness, and autogenic training are core components.
  Arms: Intervention
Other: Usual Care — Usual social and clinical services provided to patients at the recruiting clinic
  Arms: Control

SUMMARY:
Women living with HIV have 2-4x higher risk for cardiovascular disease compared to women without HIV, with women living with HIV in the Southern US being particularly at risk. While an increased prevalence of traditional risk factors (e.g., hypertension, diabetes, and obesity) partially explain this risk, evidence suggests that increased exposure to structural and social stressors (e.g., poverty, discrimination, and stigma) among women living with HIV in the South negatively contribute to cardiovascular disease disparities through their impact on stress. The Stress Management and Resiliency Training (SMART) program is an effective, evidence-based intervention proven to improve resiliency to environmental stressors and reduce the physiologic responses to stress which contribute to cardiovascular disease. While the SMART program has demonstrated efficacy in a wide range of populations and settings, it has not been designed for or tested among women living with HIV in the South, where unique cultural and faith-based context may diminish the uptake and value of the intervention to mitigate cardiovascular disease risk. The purpose of this study is to adapt the evidence-based SMART program in consideration of the needs and contexts of women living with HIV in the Southern US and pilot the adapted intervention to establish the feasibility, acceptability, and preliminary impact of the adapted intervention to reduce stress and mitigate cardiovascular disease risk among this population.

ELIGIBILITY:
Inclusion Criteria:

1. cis-gender females at least 18 years of age
2. HIV-seropositive and a patient of the recruiting clinic
3. English speaking

Exclusion Criteria:

1. severe mental illness
2. not being willing able to provide informed consent
3. not willing or able to attend study visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender women for intervention randomization
Enrollment: 48 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure at baseline, week 8, and week 20 | baseline - week 8 - week 20
  Measure blood pressure at baseline, end of intervention, and at 12-week follow-up
Change in Center for Epidemiological Studies Depression Scale Score | baseline - week 8 - week 20
  Higher score indicates more depressive symptoms (0-60 Range)
Change in Generalized Anxiety Disorder-7 Scale Score | baseline - week 8 - week 20
  Higher scores indicate greater symptoms of anxiety (0-21 Range)
Changes in Perceived Stress Scale Scores | baseline - week 8 - week 20
  Higher scores indicate greater perceived stress (0 - 40 Range)
Changes in Connor-Davidson Resilience Scale | baseline - week 8 - week 20
  Higher scores indicate greater resilience (0-100 Range)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided